CLINICAL TRIAL: NCT02542592
Title: Effect of Preoperative Intravenous High Dose Methylprednisolone on Immune Signaling in Patients Scheduled for Total Hip-arthroplasty
Brief Title: Effect of Methylprednisolone on Immune Signaling in Hip-arthroplasty Patients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Viktoria Oline Lindberg-Larsen, MD, PhD student, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: HK_VL_08_2015a; 2015-000102-19 (EudraCT Number)
Record Dates: First submitted 2015-09-03; First posted 2015-09-07 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Osteoarthrosis
Keywords: Glucocorticoids; Immune Signaling; Recovery; Hip arthroplasty, total
MeSH Terms: conditions — Osteoarthritis | interventions — Methylprednisolone; Methylprednisolone Hemisuccinate; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Methylprednisolone (Active Comparator): Preoperative single high dose of Solu-Medrol 125 mg iv.
  Interventions: Drug: Methylprednisolone
- Placebo (Placebo Comparator): Preoperative single dose of isotonic Sodium Chloride
  Interventions: Drug: Isotonic Sodium Chloride

INTERVENTIONS:
Drug: Methylprednisolone — Comparison of preoperative single high dose of Methylprednisolone 125 mg iv. and isotonic Sodium Chloride (placebo)
  Other Names: Solu-Medrol
  Arms: Methylprednisolone
Drug: Isotonic Sodium Chloride — Placebo
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
The study evaluates the pathophysiological effects of a single dose Methylprednisolone administered prior to total hip-arthroplasty (THA) surgery. The investigators examine the effect on immune signaling and recovery after surgery.

Half of participants will receive intravenous Solu-Medrol 125 mg, while the other half will receive placebo.

The investigators hypothesize that the group receiving Methylprednisolone will experience a positive modulation of the immune response and an enhanced recovery.

DETAILED DESCRIPTION:
The anti-inflammatory effects of glucocorticoids are well known. The beneficial effects on postoperative pain, postoperative nausea and vomiting are well-documented.

Hip-arthroplasty surgery and the inflammatory stress response in general affect the potential of recovery. The basic physiological mechanisms behind restoration of recovery after surgery are still unresolved. The many different immune cells involved in the complex signal response enables wound healing and recovery, and the individual immune signal pattern might be able to predict recovery. The effects of glucocorticoids on this immune signal pattern is unknown and calls for further investigation.

The study is to be considered as exploratory. This study is embedded in a primary study registrated as: NCT02445898

For further details please view the EudraCT registration:

EudraCT nr.: 2015-000102-19

ELIGIBILITY:
Inclusion Criteria:

* Osteoarthrosis
* Undergoing total unilateral hip-arthroplasty surgery
* Speak and understand Danish
* Have given informed content

Exclusion Criteria:

* Revision or bilateral hip-arthroplasty surgery
* General anaesthesia
* Allergy or intolerance towards Methylprednisolone
* Local or systemic infection
* Permanent systemic treatment with steroids within 30 days peroperatively
* Insulin-dependent diabetes
* Atrial fibrillation
* Neurological disease incl. Parkinsons
* Daily use of hypnotics or sedatives
* Alcohol abuse >35 units per week
* Active treatment of ulcer within 3 months preoperatively
* Cancer disease
* Autoimmune disease incl. rheumatoid arthritis
* Pregnant or breast feeding women
* Menopause <1 year

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2015-09; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Change in concentration of plasma-STAT3 (Signal transducer and activator of transcription) from baseline to 48 hours after surgery | 48 hours after surgery

SECONDARY OUTCOMES:
Change in concentration of plasma-STAT3 from baseline to 14 days after surgery | 14 days after surgery
Change in concentration of plasma-CREB (Adenosine 3',5'-monophosphate response element-binding protein) from baseline to 14 days after surgery | 14 days after surgery
Change in concentration of plasma-NF-kB (Nuclear factor kB) from baseline to 14 days after surgery | 14 days after surgery
Change in Surgical Recovery Scale score from baseline to 28 days after surgery | 28 days after surgery
Change in modified WOMAC (Western Ontario and McMaster Universities Arthritis Index) score from baseline to 28 days after surgery | 28 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Viktoria Lindberg-Larsen, MD, Principal Investigator — Section for Surgical Pathophysiology, Rigshospitalet
Locations (1):
- Copenhagen University Hospital, Bispebjerg, Copenhagen NV, Denmark

REFERENCES:
- [Background] Stoecklein VM, Osuka A, Lederer JA. Trauma equals danger--damage control by the immune system. J Leukoc Biol. 2012 Sep;92(3):539-51. doi: 10.1189/jlb.0212072. Epub 2012 May 31. PMID 22654121
- [Background] Wilmore DW. From Cuthbertson to fast-track surgery: 70 years of progress in reducing stress in surgical patients. Ann Surg. 2002 Nov;236(5):643-8. doi: 10.1097/00000658-200211000-00015. PMID 12409671
- [Background] Baigrie RJ, Lamont PM, Kwiatkowski D, Dallman MJ, Morris PJ. Systemic cytokine response after major surgery. Br J Surg. 1992 Aug;79(8):757-60. doi: 10.1002/bjs.1800790813. PMID 1393463
- [Background] Giannoudis PV, Smith RM, Perry SL, Windsor AJ, Dickson RA, Bellamy MC. Immediate IL-10 expression following major orthopaedic trauma: relationship to anti-inflammatory response and subsequent development of sepsis. Intensive Care Med. 2000 Aug;26(8):1076-81. doi: 10.1007/s001340051320. PMID 11030163
- [Result] Gaudilliere B, Fragiadakis GK, Bruggner RV, Nicolau M, Finck R, Tingle M, Silva J, Ganio EA, Yeh CG, Maloney WJ, Huddleston JI, Goodman SB, Davis MM, Bendall SC, Fantl WJ, Angst MS, Nolan GP. Clinical recovery from surgery correlates with single-cell immune signatures. Sci Transl Med. 2014 Sep 24;6(255):255ra131. doi: 10.1126/scitranslmed.3009701. PMID 25253674
- [Derived] Ganio EA, Stanley N, Lindberg-Larsen V, Einhaus J, Tsai AS, Verdonk F, Culos A, Ghaemi S, Rumer KK, Stelzer IA, Gaudilliere D, Tsai E, Fallahzadeh R, Choisy B, Kehlet H, Aghaeepour N, Angst MS, Gaudilliere B. Preferential inhibition of adaptive immune system dynamics by glucocorticoids in patients after acute surgical trauma. Nat Commun. 2020 Jul 27;11(1):3737. doi: 10.1038/s41467-020-17565-y. PMID 32719355